CLINICAL TRIAL: NCT06493071
Title: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) as an Anti-inflammatory Strategy for the Treatment of Depression Following Spinal Cord Injury
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) for Inflammation and Depression Following SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13842
Record Dates: First submitted 2024-06-17; First posted 2024-07-09 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-07

CONDITIONS: Spinal Cord Injury; Depression
Keywords: Vagus Nerve Stimulation; Inflammation; Kynurenine; Spinal Cord Injury; Depression
MeSH Terms: conditions — Spinal Cord Injuries; Depression; Inflammation

STUDY DESIGN:
Intervention Model Description: Eligible participants who consent to study participation will be randomized to one of two groups: active taVNS, or sham taVNS. Each group will undergo 30 days of the respective treatment.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active taVNS (Experimental): Stimulation will target the auricular branch of the vagus nerve by applying stimulation to the cymba conchae region of the ear using the NEMOS® taVNS device (taVNS Technologies, Erlangen, Germany).
  Interventions: Device: Active Transcutaneous Auricular Vagus Nerve Stimulation
- Sham taVNS (Sham Comparator): Stimulation will target the ear lobe using the NEMOS® taVNS device (taVNS Technologies, Erlangen, Germany). Stimulation will be applied to the ear lobe in order to ensure participant feel the stimulation while avoiding activation of the vagus nerve.
  Interventions: Device: Sham Transcutaneous Auricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Active Transcutaneous Auricular Vagus Nerve Stimulation — Stimulation will target the auricular branch of the vagus nerve by applying stimulation to the cymba conchae region of the ear using the tVNS R device (taVNS Technologies, Erlangen, Germany). To achieve adequate stimulation while avoiding unpleasant or painful sensations, the stimulation intensity will be gradually increased in increments of 0.1mA until the subjective pain threshold is reached, and then reduced to a stimulus intensity just below the individuals pain threshold (expected range based on prior studies 1 - 3.2mA). Pulse width will be set at 100μs and frequency will be set at 25Hz. Parameters will be set for the duration of the intervention consisting of 4 hours of daily stimulation for a period of 30 days.
  Other Names: tVNS R
  Arms: Active taVNS
Device: Sham Transcutaneous Auricular Vagus Nerve Stimulation — Stimulation will target the ear lobe using the NEMOS® taVNS device (taVNS Technologies, Erlangen, Germany). To achieve adequate stimulation while avoiding unpleasant or painful sensations, the stimulation intensity will be gradually increased in increments of 0.1mA until the subjective pain threshold is reached, and then reduced to a stimulus intensity just below the individuals pain threshold (expected range based on prior studies 1 - 3.2mA). Pulse width will be set at 100μs and frequency will be set at 25Hz. Participants will perform 4 hours of stimulation per day for a period of 30 days. Stimulation will be applied to the ear lobe in order to ensure participant feel the stimulation while avoiding activation of the vagus nerve.
  Other Names: tVNS R
  Arms: Sham taVNS

SUMMARY:
Spinal cord injury (SCI) has been shown to be associated with impairment to the autonomic nervous system in the form of reduced activity of a key nerve known as the vagus nerve. As the vagus nerve has an important role in regulating inflammation and is associated with depression, it may represent a key mechanism which contributes to chronic inflammation and depression following SCI.

A technique known as transcutaneous auricular vagus nerve stimulation (taVNS) can stimulate the vagus nerve non-invasively through an electrode applied on the skin of the ear. This technique has been shown to effectively reduce inflammation and improve symptoms of depression in other populations without any serious adverse events. However, it has not been assessed in individuals with SCI.

The primary objective of this study is to assess the efficacy of taVNS therapy for the treatment of inflammation and depression. Autonomic function as assessed by measures of heart rate variability (HRV) will also be assessed to quantify changes in vagal tone. The study will be conducted over a 2-year period, with 44 individuals with SCI and depression participating. Participants will be randomly assigned to receive either active taVNS or a placebo (sham) treatment over a 30-day period.

The researchers will assess changes in depression symptoms, autonomic function (heart rate variability), and biomarkers related to inflammation at baseline and 30-days. Safety and adherence will also be evaluated to confirm the feasibility for long-term use.

This study aims to explore a novel and non-invasive treatment strategy for depression in individuals with spinal cord injury. If taVNS is found to be safe, effective, and feasible for SCI patients, it could offer a simple, cost-effective way to address chronic inflammation and depression in this population.

DETAILED DESCRIPTION:
Depression and chronic inflammation are highly prevalent following SCI Inflammation plays an increasingly appreciated role in the pathology of depression. One key mechanism is the ability to dysregulate a key metabolic pathway (the Kynurenine pathway) resulting in serotonin deficits and increased production of neurotoxic metabolites. Prior research from our lab has demonstrated the efficacy of diet and exercise to affect this pathway and improve clinical symptoms. However, we have shown that the burdensome nature of such interventions limits long-term adherence in SCI. Stimulating the vagus nerve has been shown to induce anti-inflammatory effects in populations with chronic inflammation (e.g. rheumatoid arthritis; Crohn's disease) and lower scores of depression.

However, the potential benefits of a chronic vagus nerve stimulation intervention has not been assessed in individuals with SCI. Transcutaneous auricular vagus nerve stimulation (taVNS) is a simple to administer and non-invasive neurostimulatory technique which can stimulate the vagus nerve via the skin of the ear. Given that SCI is associated with chronic inflammation, high rates of depression, and reductions in vagal tone, they may represent a population that would be particularly susceptible to the benefits of this low-burden, low-cost treatment strategy.

The overall objective of this study is to demonstrate that transcutaneous auricular vagus nerve stimulation (taVNS) therapy is a safe and feasible treatment which effectively activates the vagus nerve in individuals with SCI. The study will also provide preliminary efficacy data related to the impact on symptoms of depression and inflammatory biomarkers.

Participants will be randomized to receive either active taVNS therapy (treatment group), or sham taVNS therapy (placebo group). The intervention will be performed over a 30-day period and will follow the recommended daily stimulation of 4-hours per day with at least 1-hour carried out continuously (for a total of 30 sessions).

All participants will have an in-person baseline visit to determine optimal taVNS stimulation parameters and be trained on instructions for use. For the active stimulation group, stimulation will target the auricular branch of the vagus nerve by applying stimulation to the cymba conchae region of the left ear using the tVNS R device (taVNS Technologies, Erlangen, Germany). For the sham group, stimulation will target the earlobe, which will allow the participant to feel the stimulation, while avoiding stimulation of the auricular branch of the vagus nerve. To achieve adequate stimulation while avoiding unpleasant or painful sensations, the stimulation intensity will be gradually increased in increments of 0.1mA until the subjective pain threshold is reached, and then reduced to a stimulus intensity just below the individuals pain threshold (expected range based on prior studies 1 - 3.2mA). Pulse width will be set at 100μs and frequency will be set at 25Hz as performed in our previous protocol in spinal cord injured patients (approved by Health Canada: 364351 and shown to safely and effectively increase vagal tone). The stimulation parameters determined during this in-person baseline visit will be locked for the duration of the 30-day intervention.

Upon establishing appropriate stimulation parameters, each participant will be trained on instructions for use. As the tVNS R device is designed to be carried out independently by the patient, instructions for use are simple and user friendly. The participant will be instructed to: 1) clean the ear using provided alcohol swabs, 2) place the electrode in the ear in the appropriate orientation (depending on group allocation), 3) turn the device on by pressing the 'ON' button, and 4) begin stimulation by pressing the 'START/STOP button once. Participants may then place the device in their pocket and go about their daily activities as normal. The device will display percent completion of the daily 4-hour stimulation period so that participants are aware of there daily progress and when the session is complete.

At the initial study visit, as well as the 30-day post study visit, participants will also undergo an assessment of heart rate variability (HRV), depression, and inflammatory biomarkers:

HRV will be assessed via electrocardiogram (ECG) to assess changes in autonomic function related to vagal tone. For the collection of ECG signals participants will be instructed to avoid caffeine, alcohol, and strenuous exercise for at least 24 hours prior to assessment. Participants will be instructed to remain relaxed, focus on breathing, and avoid speaking throughout the protocol. ECG recording will be collected using the Polar H10 heart monitor. Continuous heart rate will be recorded for a period of 5-minutes to obtain a baseline measure. This process will be repeated following the 30-day intervention period at the post testing session. ECG data will be imported to Kubios software for analysis of root mean square of successive differences (RMSSD) as well as high frequency (HF) power. RMSSD is a time domain measure of heart rate variability corresponding to the variability in the intervals between successive heartbeats and is a measure of vagal tone. HF power is a frequency domain measure of heart rate variability corresponding to heart rate fluctuations occurring in the frequency range of 0.15 to 0.4Hz and also reflects vagal tone. RMSSD (which is less influenced by breathing rate) will be the primary assessment of vagal tone, and HF power will be assessed to ensure consistency in measures. Measures of vagal tone will be assessed at baseline and post-intervention to assess whether the intervention successfully targets the vagus nerve and increases vagal tone.

Depression will be assessed via the Patient Health Questionnaire (PHQ-9) at baseline, and 30-days (post-intervention). The PHQ-9 has been shown to be a valid assessment for major depressive disorder in individuals with SCI. The PHQ-9 is a 9-item questionnaire with items pertaining to feelings over the previous 2-weeks. Each item is scored on a scale from 0 ("not at all") to 3 ("nearly every day") with total scores allowing for assessment of depression severity. A score ranging from 0-4 suggests "none-minimal" depression severity, 5-9 suggests mild depression severity, 10-14 suggests moderate depression severity, 15-19 suggests moderately severe depression severity, and 20-27 suggests severe depression severity. The instrument also includes a functional health assessment which asks participants how emotional difficulties or problems impact work, life at home, or relationships with other people with responses ranging from "not difficult at all" to "extremely difficult". A PHQ-9 score ≥ 10 has a sensitivity of 88% and a specificity of 88% for major depression. The PHQ-9 will be assessed at baseline, post-intervention and weekly throughout the intervention.

Biomarkers will be assessed via blood samples (20 ml) collected by a certified phlebotomist for the quantification of plasma biomarkers. Blood draws will be performed at baseline, and post-intervention. Plasma concentrations of the pro-inflammatory cytokines tumour necrosis factor-alpha (TNF-α), C-reactive protein (CRP), interleukin-6 (IL-6), interleukin-1 beta (IL-1β), and interferon-gamma (IFN-y) will be quantified using 32x4 simple plex multianalyte cartridge for the Ella automated immunoassay system (ProteinSimple, San Jose, California). Each of the cytokines TNF-α, IL-1β, IL-6, and IFN-y have been shown to dysregulate the KYN pathway, while CRP is a ubiquitous measure of inflammation. Plasma concentrations of metabolites of the kynurenine pathway including tryptophan (TRP), kynurenine (KYN), kynurenic acid (KYNA), and quinolinic acid (QUIN) will be quantified in triplicate via enzyme-linked immunosorbent assay (ImmuSmol, Pessac, France).

In addition safety and adherence will be monitored throughout the intervention period via twice weekly phone calls. Any incidence of treatment-emergent adverse events during the intervention will be recorded each week and compared between the taVNS and control groups. A description of the adverse event, number of events, and total number of participants affected will be recorded. Adherence will be assessed each week by the number of days whereby participants completed the full 4-hour session. These phone calls will include completion of the PHQ-9 to monitor for any signs of worsening depression.

ELIGIBILITY:
Inclusion criteria:

1. SCI of any level or severity
2. 18 years of age or older
3. scores suggesting mild - moderately severe depression on the PHQ-9 (5 - 19)
4. stable dose of depression medications

Exclusion criteria:

1. Prone to autonomic dysreflexia
2. Severe depression as assessed by PHQ-9 (≥20)
3. Suicidal ideation
4. presence of cardiovascular disease
5. pacemaker or other implanted electrical device (e.g. cochlear implant, implanted vagus nerve stimulator, cardiac pacemaker)
6. people with cerebral shunts
7. people with epilepsy
8. people who pregnant or attempting to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events During Intervention | 30 days
  All adverse events which occur during the intervention will be recorded during the twice weekly phone calls and/or study visits and compared between the active taVNS and sham taVNS conditions. A description of the adverse event, number of events, and total number of participants affected will be recorded.
Change in Root Mean Square of Successive Differences (RMSSD) | 30 days
  HRV will be assessed via electrocardiogram (ECG) to assess changes in autonomic function related to vagal tone. Continuous heart rate will be recorded at rest for a period of 5-minutes to obtain a baseline measure. This process will be repeated following the 30-day intervention period at the post testing session. ECG data will be used for analysis of root mean square of successive differences (RMSSD). RMSSD will be assessed at baseline and post-intervention to assess whether the intervention successfully targets the vagus nerve and increases vagal tone.

SECONDARY OUTCOMES:
Change in High Frequency (HF) Power | 30 days
  Changes in autonomic function related to vagal tone will also be assessed via changes in high frequency (HF) power to confirm changes seen in root mean square of successive differences (RMSSD). HRV will be assessed via electrocardiogram (ECG). Continuous heart rate will be recorded at rest for a period of 5-minutes to obtain a baseline measure. This process will be repeated following the 30-day intervention period at the post testing session. ECG data will be used for analysis of HF power. HF Power will be assessed at baseline and post-intervention to assess whether the intervention successfully targets the vagus nerve and increases vagal tone.
Change in Symptoms of Depression | 30 days
  Depression will be assessed via the Patient Health Questionnaire (PHQ-9) at baseline, and 30-days (post-intervention). The PHQ-9 has been shown to be a valid assessment for major depressive disorder in individuals with SCI. The PHQ-9 is a 9-item questionnaire with items pertaining to feelings over the previous 2-weeks. Each item is scored on a scale from 0 ("not at all") to 3 ("nearly every day") with total scores allowing for assessment of depression severity. A score ranging from 0-4 suggests "none-minimal" depression severity, 5-9 suggests mild depression severity, 10-14 suggests moderate depression severity, 15-19 suggests moderately severe depression severity, and 20-27 suggests severe depression severity. A PHQ-9 score ≥ 10 has a sensitivity of 88% and a specificity of 88% for major depression.
Change in Plasma Cytokines | 30 Days
  Blood samples (20 ml) will be collected by a certified phlebotomist at baseline and 30-days (post intervention) for the quantification of plasma cytokines (pg/ml). Plasma concentrations of the pro-inflammatory cytokines tumour necrosis factor-alpha (TNF-α), C-reactive protein (CRP), interleukin-6 (IL-6), interleukin-1 beta (IL-1β), and interferon-gamma (IFN-y) will be quantified using 32x4 simple plex multianalyte cartridge for the Ella automated immunoassay system (ProteinSimple, San Jose, California). Each of the cytokines TNF-α, IL-1β, IL-6, and IFN-y have been shown to dysregulate the KYN pathway, while CRP is a ubiquitous measure of inflammation.
Change in Plasma Kynurenines | 30 days
  Blood samples (20 ml) will be collected by a certified phlebotomist at baseline and 30-days (post intervention) for the quantification of plasma kynurenines (ng/ml). Plasma concentrations of the kynurenines tryptophan (TRP), kynurenine (KYN), kynurenic acid (KYNA), and quinolinic acid (QUIN) will be quantified in triplicate via enzyme-linked immunosorbent assay (ImmuSmol, Pessac, France).
Program Adherence Rates | 30 Days
  Adherence will be assessed each week by the number of days whereby participants completed the full 4-hour session.

CONTACTS AND LOCATIONS:
Overall Officials: David J Allison, PhD., Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Parkwood Institute, St Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No